CLINICAL TRIAL: NCT05510193
Title: Redesign, Implementation and Evaluation of the Effectiveness of the Aktio Myoelectric Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Antioquia (Other)
Collaborators: Hospital San Vicente Fundación (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-30970
Record Dates: First submitted 2022-06-28; First posted 2022-08-22 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-10

CONDITIONS: Upper Limb Amputation Below Elbow (Injury); Prosthesis User; Satisfaction, Patient
Keywords: Myoelectric prosthesis; 3D printing
MeSH Terms: conditions — Wounds and Injuries; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aktio (Experimental): Use of the prosthesis for 2 weeks, after a 3-session training
  Interventions: Device: Aktio prosthesis
- Control (No Intervention): Non-use of the prosthesis

INTERVENTIONS:
Device: Aktio prosthesis — Transradial myoelectric prosthesis
  Arms: Aktio

SUMMARY:
In Latin America, Colombia ranks fourth in countries with the highest number of people with disabilities (6.4%), 80% of whom live in low socioeconomic strata, have little access to education and high unemployment rates. Of these nearly 3 million people with this condition, an estimated 11,476 need upper limb prostheses, 12% of whom have transradial or below-elbow amputation. Although many of the functions that have been lost by amputation can be recovered with a prosthesis, few people in Colombia use these devices. This is because, currently, only aesthetic and mechanical options are found, and the most advanced options, such as myoelectric ones, are manufactured in other countries, have very high prices and are not designed according to local needs. The only option manufactured at the national level is the one developed by Protesis Avanzadas S.A.S., but it still has aspects to improve that would lead it to better adapt to the needs of Colombian users.

All of the above shows the evident need for the country to generate products that can help this population. The objective of this project is then to redesign, implement and evaluate the effectiveness of a good quality transradial myoelectric prosthesis, focused on the Colombian amputee population and improving acceptance rates. For the design phase of the study, a group made up of health professionals and patients with transradial amputation will be included to evaluate the preferences and priorities of their prosthesis. For pre-commercial validation, an effectiveness study will be carried out by means of a randomized crossover clinical trial with 12 participants in which the functioning and quality of life of the user with and without the prosthesis and satisfaction with it will be analyzed using methods of Bayesian statistics. This study is expected not only to improve the quality of life of people with transradial amputation and their families, but also to provide a functional option for the health system.

DETAILED DESCRIPTION:
Methodology and work plan of the pre-commercial validation process The methodology for the redesign of the transradial myoelectric prosthesis will seek to add value to the current design, by increasing the value perceived by the buyer by providing additional attributes to the current ones. The methodology will be divided into five main phases that go from the clarification of the objectives that are expected to be satisfied with the design, to the creation and evaluation of a functional prototype that has been improved after carrying out performance tests, and carrying out an evaluation. of effectiveness, in addition to a parallel phase to all that includes the financial analysis. The details of each of the phases are found below.

Conceptual design During this phase, we will seek to define the concept on which the redesign of the transradial prosthesis will be developed based on the Cross Design Method. Initially, a complete and clear approach must be made of the objectives that the prosthesis must satisfy through the clarification of objectives. Then, we will continue with the establishment of functions. Starting from the identification of the level of generality or detail at which to work, the functions and limits of the problem to be solved will be defined, establishing the specific functions that the prosthesis must satisfy, regardless of the physical components that could be used.

Subsequently, the requirements will be set, where the performance specification of the prosthesis will be defined, which will allow evaluating that the proposed solutions are within acceptable limits. In addition, the determination of characteristics will be elaborated, where the desirable attributes of the new product will be compared - from the customer's point of view - with the previously defined engineering requirements. This comparison will be made through the deployment of the quality function, which implies interviews or surveys with possible users and experts on the subject, group sessions, search for the state of the art, among others.

Finally, the generation of alternatives and their evaluation will be carried out. The generation of alternatives is based on the morphological diagram method, which presents the full range of elements, components or secondary solutions that can be combined to form different solutions, from which the alternative designs will be defined. During the evaluation of alternatives, the different alternative designs will be evaluated according to the previously defined requirements and objectives.

For these activities, there will be a group of participants with transradial amputation who agree to enter the study. In the session, the priorities and preferences of patients regarding the use of prostheses and the needs that these should cover will be qualitatively evaluated. It will investigate aspects such as usability, comfort, adaptation, strength, mobility, performance in activities of daily living and quality of life.

Additionally, the participation of professionals involved in the rehabilitation of patients with upper limb amputation will be sought, who will also be interviewed to define the objectives and clinical aspects to be taken into account in the design of the prosthesis. Likewise, both entities (Prótesis Avanzadas and the University of Antioquia) will keep the deliverables of this design phase.

Materialization design This design phase follows the methodology established for Engineering Design by Pahl and Beitz, and in it the design of the transradial myoelectric prosthesis is developed from the concept defined in the previous phase and considering the technical and economic criteria of the same. In addition, it must lead to the definitive design of the prostheses, after verifying that the function, durability, production, assembly, operation and costs of the design meet the specifications.

It is important to keep in mind that due to the complexity of materialization design (i.e. some activities must be repeated when more information is available, changes made in one area of the design may affect others, several actions must be carried out simultaneously), particular problems that are found can generate deviations from what was planned. Therefore, it is recommended to develop this phase starting from the most general to the most specific and defining verification points to make corrections.

Both entities will retain the deliverables from this design phase. Detail design In this phase of the design, it is expected to obtain the necessary documents to produce myoelectric prostheses. In our specific case, since the Prosthetics Advanced production system is based on 3D printing, the main documents will be the CAD files of the designed components, the list of parts that includes both the commercial elements and the printed components, the assembly drawing and the manual of use of the prosthesis. Both entities will retain the deliverables from this design phase.

Pre-commercial evaluation As a final phase of the design, a prototype will be manufactured, and performance tests will be carried out. Likewise, production tests will be carried out in which problems with the creation of the prostheses are identified. Finally, with the results of the tests, the design improvements will be developed, updating the necessary documents to produce the prostheses and obtaining a prototype of the improved design. Once the design has been defined, an effectiveness study will be carried out with patients with transradial amputation.

Design of the effectiveness study A clinical trial with a randomized crossover design will be carried out to define the moment of the intervention in twelve participants. This type of design reduces the influence of confounding variables because subjects can act as their own control in the trial and is ideal for evaluating interventions in chronic and stable conditions, such as limb amputations.

The intervention will then be compared, that is, the use of the myoelectric prosthesis versus the non-use of the prosthesis. It is assumed that there is no "carryover" effect as the intervention (prosthesis) is expected to have the desired effect while in use and not have a residual effect on function upon removal, therefore no washout period is required between removal. the interventions.

Selection and sample size Sampling will be done for convenience and patients will be selected from the physiatry, plastic surgery or orthopedics clinic of the participating institutions. The number of patients was selected considering the costs of the design, the costs and time required for the elaboration of the prostheses, the time required for effectiveness tests and the resources available for the project.

Intervention and control Each prosthesis will be delivered by members of the design team and a physical or occupational therapist, who will make the necessary adjustments for adaptation and will train in its use during two sessions of 3 hours each. In the intervention group, the patients will use the prosthesis for a period of two weeks and after this time they will be scheduled for the application of the functioning, satisfaction and quality of life scales. The patients assigned to the control group will be cited for the application of the functioning and quality of life scales. The controls will be carried out without the use of the prosthesis since this is the most common scenario in upper limb amputees and we want to demonstrate that the use of prostheses is superior to "no treatment".

No washout period is required between periods as the intervention (prosthesis) is expected to have the desired effect while in use and not have a residual effect upon removal. Blinding of participants or investigators will not be possible due to the type of intervention and outcome measurement.

Outcomes For this study, selected outcomes will be evaluated: functioning defined as performance in daily activities, both self-reported and observed; satisfaction with the prosthesis and health-related quality of life. Recently, the Working Group on Upper Extremity Prosthetic Outcome Measures (ULPOM) recommended the use of the World Health Organization International Classification of Functioning, Disability and Health (ICF) as the ideal framework for selecting instruments and outcomes, and highlighted the importance of selecting assessment tools that take into account each of the important elements of the ICF, including body structures and functions (prosthesis performance), activity (performing tasks), and participation (use of the device). prosthetics in real life situations).

Data collection plan To obtain the data of the possible participants, patients who meet the inclusion criteria will be contacted, invitations to be part of the study will be sent, with a summary of the study, and visits will be planned after making appointments with those who have agreed to participate. During the visits, compliance with the inclusion criteria will be confirmed, the objectives and methodology of the project will be explained, and informed consent will be obtained. The data will be taken from primary sources through the application of instruments completed by the participant and performance instruments supervised by one of the researchers. The random allocation will be made using computer-generated codes, in sealed and opaque envelopes. Two measurements of the outcomes will be made, with and without the use of prostheses, separated by a period of 2 weeks. One person will be responsible for data collection and should verify the quality of the records and the presence of missing data before leaving the participant's side. The principal investigator will review the quality of the records and the presence of missing data that would require recontacting the participant in person or by phone.

The data obtained through the application of the instruments will be digitized by one of the researchers and reviewed by the principal investigator to control the quality of the data. Everything will be recorded in a database in MS Access®.

Ethical considerations According to Resolution 8430 of 1993, which establishes the scientific, technical, and administrative standards for health research, it is considered low-risk research. Approval from a Human Research Bioethics Committee will be sought.

Research involving human beings must be governed by three basic ethical principles. The principle of respect for people, which refers to autonomy in participating in a study; it is guaranteed through informed consent and respect for autonomy, clarifying that participation is voluntary and can be stopped at any time during the study. The principle of beneficence refers to the effort to promote the well-being of the research subject, seeking to achieve the maximum benefit with the minimum risk and harm. The principle of justice is related to the equitable selection of participants and equitable access to risks and benefits.

The research team is committed to complying with the standards of good clinical practice in research. We will provide detailed information to each participant about the purpose and importance of the study and request informed consent from each one. The research team will be responsible for the confidentiality of patient data. The information will be encrypted and kept in custody. Upon completion of the investigation, the team agrees to disclose the results.

It should be noted that prostheses are classified as non-invasive medical devices and that the Prótesis Avanzadas company has experience in the production of 3D-printed prostheses for upper limbs.

ELIGIBILITY:
Inclusion Criteria:

* Who live in Medellín or the metropolitan area and can travel to the place of evaluation.
* Patients who are able to understand and follow orders.

Exclusion Criteria:

* Patients with bilateral upper limb amputation.
* Patients with skin or soft tissue injuries that contraindicate the use of prostheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-27 (Estimated)

PRIMARY OUTCOMES:
Functional status | 2 weeks after training with the prostheses in the intervention group
  Auto-reported functioning. Measured with the Orthotics and Prosthetics Users Survey - Upper extremity Functional status (OPUS - UEFS). It is an instrument to report the difficulty or ease in the execution of 23 tasks of daily life and self-care. Tasks are rated on a 1-5 point scale (very easy to unable to do the activity), regardless of how the activities are performed (with or without a prosthesis). Scores range from 0 to 100, with higher scores indicating more difficulty in performing activities.

SECONDARY OUTCOMES:
Observed performance | 2 weeks after training with the prostheses in the intervention group
  Observed performance. Measured with the Brief activity performance measure for upper limb amputees (BAM-ULA). It is an observational measure of activity performance. Each item is scored from zero for "cannot complete" or one for "completed". The scores for each item are added together to get the overall completion score for the task. Summary scores are calculated only when all ten items are scored. Higher scores on activity completion indicate better performance.
Satisfaction with prosthesis | 2 weeks after training with the prostheses in the intervention group
  Satisfaction with prosthesis. Measured with the Prosthetics Users Survey - Satisfaction (OPUS Satisfaction)
Quality of life related to health and prosthesis use | 2 weeks after training with the prostheses in the intervention group
  Perceived quality of life related to health and prosthesis use. Measured with the Orthotics and Prosthetics Users Survey - Health Quality of Life Index (OPUS - QoL). The OPUS Health Quality of Life Score consists of 23 items that assess health-related quality of life. Items are rated on a 5-point rating scale. The total instrument score is calculated by adding the scores of the 23 items. A higher score indicates a better result.

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Lemos, Principal Investigator — Universidad de Antioquia
Locations (2):
- Colombia (2):
  - Hospital San Vicente Fundación, Medellín, Antioquia
  - Prótesis Avanzadas S.A.S, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: Yes
Databases with results of scores in questionnaires
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available once it is finished collecting in the 12 participants. There will be no time limit for its availability.
Access Criteria: They will be shared at the request of the interested parties, who establish a clear objective for the use of the data in the request.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05510193/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT05510193/ICF_001.pdf